CLINICAL TRIAL: NCT00763451
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, 24-week Study Followed by an Extension Assessing the Efficacy and Safety of AVE0010 in Two Titration Regimens on Top of Metformin in Patients With Type 2 Diabetes Not Adequately Controlled With Metformin
Brief Title: GLP-1 Receptor Agonist Lixisenatide in Patients With Type 2 Diabetes for Glycemic Control and Safety Evaluation, on Top of Metformin
Acronym: GETGOAL-F1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC10743; 2008-001002-16 (EudraCT Number)
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: hyperglycemia, GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — lixisenatide; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lixisenatide (Two-Step Titration) (Experimental): 2-step initiation regimen of lixisenatide: 10 microgram (mcg) once daily (QD) for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector; Drug: Metformin
- Lixisenatide (One-Step Titration) (Experimental): 1-step initiation regimen of lixisenatide: 10 mcg QD for 2 weeks, then 20 mcg QD up to the end of treatment.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector; Drug: Metformin
- Placebo (Two-Step Titration) (Placebo Comparator): 2-step initiation regimen of volume matching placebo: 10 mcg QD for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
  Interventions: Drug: Placebo; Device: Pen auto-injector; Drug: Metformin
- Placebo (One-Step Titration) (Placebo Comparator): 1-step initiation regimen of volume matching placebo: 10 mcg QD for 2 weeks, then 20 mcg QD up to the end of treatment.
  Interventions: Drug: Placebo; Device: Pen auto-injector; Drug: Metformin

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Self-administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Lixisenatide (One-Step Titration); Lixisenatide (Two-Step Titration)
Drug: Placebo — Self-administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Placebo (One-Step Titration); Placebo (Two-Step Titration)
Device: Pen auto-injector
  Other Names: OptiClik®
Drug: Metformin — Metformin to be continued at stable dose (at least 1.5 gram per day) up to the end of treatment.

SUMMARY:
The purpose of this study is to evaluate the benefits and risks of lixisenatide (AVE0010), in comparison to placebo, as an add-on treatment to metformin, over a period of 24 weeks of treatment, followed by an extension.

The primary objective is to assess the effects of lixisenatide when added to metformin on glycemic control in terms of glycosylated hemoglobin (HbA1c) reduction when it is used in two steps dose titration regimen at Week 24.

Secondary objectives are to assess the effects of lixisenatide when added to metformin on glycemic control in comparison to placebo in terms of HbA1c reduction when it is used in a one-step dose titration regimen, the percentage of patients with HbA1c less than 7 percent or less than or equal to 6.5%, body weight, fasting plasma glucose (FPG); to assess the safety, tolerability, pharmacokinetics (PK) and anti-lixisenatide antibody development.

DETAILED DESCRIPTION:
Patients who complete the 24-week main double-blind treatment would undergo a variable double-blind extension treatment, which ends for all patients at approximately the scheduled date of Week 76 visit (Visit 25) for the last randomized patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, diagnosed for at least 1 year at the time of screening visit, insufficiently controlled with metformin at a stable dose of at least 1.5 gram/day for at least 3 months prior to screening visit

Exclusion Criteria:

* HbA1c less than (<) 7% or greater than (>) 10% at screening
* At the time of screening age <legal age of majority
* Pregnant or breastfeeding women or women of childbearing potential with no effective contraceptive method
* Type 1 diabetes mellitus
* Treatment with an antidiabetic pharmacological agent other than metformin within the 3 months preceding the screening
* FPG at screening >250 milligram per deciliter (mg/dL) (>13.9 millimole per liter [mmol/L])
* Body mass index less than or equal to (<)20 kilogram per square meter (kg/m^2)
* Weight change of more than 5 kg during the 3 months preceding the screening visit
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease
* History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening
* Hemoglobinopathy or hemolytic anemia, receipt of blood or plasma products within 3 months prior to the time of screening
* Within the last 6 months prior to screening: history of myocardial infarction, stroke, or heart failure requiring hospitalization
* Known history of drug or alcohol abuse within 6 months prior to the time of screening
* Cardiovascular, hepatic, neurological, endocrine disease, active malignant tumor or other major systemic disease or patients with short life expectancy making implementation of the protocol or interpretation of the study results difficult, history or presence of clinically significant diabetic retinopathy, history or presence of macular edema likely to require laser treatment within the study period
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting supine systolic or diastolic blood pressure >180 millimeter of mercury (mmHg) or >95 mmHg, respectively
* Laboratory findings at the time of screening: aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase (ALP): >2 times upper limit of the normal (ULN) laboratory range; amylase and/or lipase: >3 times ULN; total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome); hemoglobin <11 gram/deciliter and/or neutrophils <1500 per cubic millimeter (mm^3) and/or platelets <100000/mm^3; positive test for Hepatitis B surface antigen (HBsAg) and/or Hepatitis C antibody (HCAb) and positive serum pregnancy test in females of childbearing potential
* Any clinically significant abnormality identified on physical examination, laboratory tests, electrocardiogram (ECG) or vital signs at the time of screening that in the judgment of the investigator or any sub-investigator precludes safe completion of the study or constrains efficacy assessment
* Patients who are considered by the investigator or any sub-investigator as inappropriate for this study for any reason (for example, impossibility to meet specific protocol requirements, such as scheduled visits, being able to do self-injections), likelihood of requiring treatment during the screening phase and treatment phase with drugs not permitted by the clinical study protocol; investigator or any sub-investigator, pharmacist, study coordinator, other study staff or relative thereof directly involved in the conduct of the protocol)
* Use of oral or injectable antidiabetic or hypoglycemic agents other than metformin (for example, sulfonylurea, alpha glucosidase inhibitor, thiazolidinedione, rimonabant, exenatide, dipeptidylpeptidase-4 (DPP-IV) inhibitor, insulin) within 3 months prior to the time of screening
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for one week or more within 3 months prior to the time of screening
* Use of any investigational drug within 3 months prior to study
* Any previous treatment with lixisenatide or participation in any previous study with lixisenatide
* Renal impairment defined with creatinine >1.4 mg/dL in women and creatinine >1.5 mg/dL in men
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including, but not limited to gastroparesis and gastroesophageal reflux disease requiring medical treatment, within 6 months prior to the time of screening
* Allergic reaction to any glucagon like peptide-1 (GLP-1) agonist in the past (for example, exenatide, liraglutide) or to metacresol
* Additional exclusion criteria at the end of the run-in phase: informed consent withdrawal; lack of compliance during the single-blind placebo run-in phase (>2 injections missed); and patient with any adverse event which precludes the inclusion in the study, as assessed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Vilnius, Lithuania
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Brastislava, Slovakia
- Sanofi-Aventis Administrative Office, Kiev, Ukraine

REFERENCES:
- [Result] Bolli GB, Munteanu M, Dotsenko S, Niemoeller E, Boka G, Wu Y, Hanefeld M. Efficacy and safety of lixisenatide once daily vs. placebo in people with Type 2 diabetes insufficiently controlled on metformin (GetGoal-F1). Diabet Med. 2014 Feb;31(2):176-84. doi: 10.1111/dme.12328. Epub 2013 Oct 24. PMID 24117597
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Ambery P, Donner TW, Biswas N, Donaldson J, Parkin J, Dayan CM. Efficacy and safety of low-dose otelixizumab anti-CD3 monoclonal antibody in preserving C-peptide secretion in adolescent type 1 diabetes: DEFEND-2, a randomized, placebo-controlled, double-blind, multi-centre study. Diabet Med. 2014 Apr;31(4):399-402. doi: 10.1111/dme.12361. Epub 2013 Dec 6. PMID 24236828

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 75 centers in 15 countries between September 29, 2008 and January 27, 2011. The overall duration of treatment was at least 76 weeks (24 weeks main double-blind treatment; variable double-blind extension treatment).
Pre-assignment Details: A total of 884 patients were screened of which 400 (45.2%) were screen failures; main reason for screen failure was glycosylated hemoglobin (HbA1c) values being out of the defined protocol range (greater than or equal to 7 percent [%] and less than or equal to 10%). A total of 484 patients were randomized.
Groups:
- Placebo (Two-Step Titration): 2-step initiation regimen of volume matching placebo: 10 microgram (mcg) once daily (QD) subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
- Placebo (One-Step Titration): 1-step initiation regimen of volume matching placebo: 10 mcg QD subcutaneously for 2 weeks, then 20 mcg QD up to the end of treatment.
- Lixisenatide (Two-Step Titration): 2-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
- Lixisenatide (One-Step Titration): 1-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 2 weeks, then 20 mcg QD up to the end of treatment.
Period: Overall Study
Arm/Group | Placebo (Two-Step Titration) | Placebo (One-Step Titration) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Started | 80 (Randomized.) | 82 | 161 | 161
Treated/Safety Population | 79 (All patients who were exposed to at least 1 dose, regardless of amount of treatment administered.) | 81 | 161 | 161
Modified Intent-to-Treat(mITT)Population | 79 (All patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment.) | 80 | 160 | 160
Completed | 67 | 60 | 121 | 131
Not Completed | 13 | 22 | 40 | 30
Not completed — Adverse Event | 4 | 6 | 19 | 14
Not completed — Lack of Efficacy | 1 | 4 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 6 | 9 | 7
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Poor Compliance to Protocol | 1 | 1 | 2 | 2
Not completed — Familial and Personal Reasons | 5 | 3 | 5 | 4
Not completed — Randomized but not Treated | 1 | 1 | 0 | 0
Not completed — Study Site Reason | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Two-step Titration) | Placebo (One-step Titration) | Lixisenatide (Two-step Titration) | Lixisenatide (One-step Titration) | Total
Number analyzed (Participants) | 79 | 81 | 161 | 161 | 482
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (8.8) | 57.5 (10.8) | 54.6 (8.9) | 55.4 (8.9) | 56.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 45 | 89 | 90 | 267
  Male | 36 | 36 | 72 | 71 | 215
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Caucasian/White | 72 | 76 | 146 | 141 | 435
  Race: Black | 0 | 1 | 2 | 1 | 4
  Race: Asian/Oriental | 5 | 4 | 11 | 13 | 33
  Race: Other | 2 | 0 | 2 | 6 | 10
  Ethnicity: Hispanic | 24 | 22 | 55 | 44 | 145
  Ethnicity: Non Hispanic | 55 | 59 | 106 | 117 | 337
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 8.03 (0.81) | 8.02 (0.84) | 8.10 (0.88) | 7.99 (0.87) | 8.04 (0.86)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] | 9.60 (2.06) | 9.31 (1.82) | 9.54 (2.50) | 9.56 (2.02) | 9.52 (2.17)
Body Weight [Mean (Standard Deviation); unit: kilogram] | 87.45 (16.32) | 88.28 (18.43) | 87.41 (16.90) | 90.21 (18.95) | 88.50 (17.77)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 6.68 (5.33) | 5.77 (4.00) | 6.01 (4.60) | 5.77 (3.85) | 6.00 (4.40)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI was calculated by dividing body weight (kilogram) by the height (meter) squared.
  kilogram per square meter (kg/m^2) | 32.38 (5.04) | 32.35 (5.86) | 32.06 (4.84) | 32.99 (5.80) | 32.47 (5.38)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: Absolute change = HbA1c value at Week 24 minus HbA1c value at baseline. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
  The "Placebo (Two-step Titration)" and "Placebo (One-step Titration)" Arms/Groups were combined as pre-specified in the study protocol
Time Frame: Baseline, Week 24
Population: mITT population:all randomized patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment, irrespective of compliance with study protocol/procedures. Last observation carried forward used. Number of patients analyzed=patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Groups:
- Placebo (Combined): Included all patients who received 2-step initiation regimen of volume matching placebo and 1-step initiation regimen of volume matching placebo.
- Lixisenatide (Two-Step Titration): 2-step initiation regimen of lixisenatide.
- Lixisenatide (One-Step Titration): 1-step initiation regimen of lixisenatide.
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 158 | 152 | 156
percentage of hemoglobin | -0.42 (0.099) | -0.83 (0.099) | -0.92 (0.101)
Statistical Analysis 1: Comparison: Placebo (Combined) vs Lixisenatide (Two-Step Titration); To detect a difference of 0.5% (or 0.4%) in absolute change from baseline in HbA1c at Week 24 between 1 lixisenatide arm and placebo (combined), 150 patients per group would provide a power of 91% (or 75%) assuming common standard deviation of 1.3% with 2-sided test at 5% significance level. Analysis of co-variance (ANCOVA) included treatment arms, randomization strata of screening HbA1c (<8.0,>=8.0%) and screening BMI (<30,>=30 kg/m^2), country as fixed effects, baseline HbA1c as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — Stepwise testing procedure applied to control type 1 error: Lixisenatide (2-step titration) was compared with Placebo (combined), if found statistically significant, then Lixisenatide (1-step titration) arm compared with Placebo (combined); Threshold for significance at 0,05 level; Least squares (LS) mean difference = -0.41, 95% CI 2-sided [-0.583 to -0.232], Standard Error of Mean 0.089
Statistical Analysis 2: Comparison: Placebo (Combined) vs Lixisenatide (One-Step Titration); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Threshold for significance at 0,05 level; Least squares (LS) mean difference = -0.49, 95% CI 2-sided [-0.670 to -0.317], Standard Error of Mean 0.090

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 1 day after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using last observation carried forward (LOCF). Here, number of patients analyzed = patients with baseline and at least 1 post-baseline FPG assessment during on-treatment period.The "Placebo (Two-step Titration)"and"Placebo (One-step Titration)"Arms/Groups were combined as pre-specified in the study protocol
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 158 | 160 | 158
mmol/L | 0.11 (0.209) | -0.56 (0.208) | -0.53 (0.212)

3. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.The "Placebo (Two-step Titration)" and "Placebo (One-step Titration)" Arms/Groups were combined as pre-specified in the study protocol
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 158 | 155 | 158
kilogram | -1.63 (0.385) | -2.68 (0.385) | -2.63 (0.389)

4. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than 7% at Week 24
Description: The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.The "Placebo (Two-step Titration)" and "Placebo (One-step Titration)" Arms/Groups were combined as pre-specified in the study protocol
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 158 | 152 | 156
percentage of participants | 24.1 | 42.1 | 47.4

5. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than or Equal to 6.5% at Week 24
Description: as for outcome 4
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 158 | 152 | 156
percentage of participants | 7.6 | 20.4 | 25.6

6. Secondary Outcome: Percentage of Patients Requiring Rescue Therapy During Main 24-Week Period
Description: Routine fasting self-measured plasma glucose (SMPG) and central laboratory FPG (and HbA1c after week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after week 12) were performed. Threshold values - from baseline to Week 8: fasting SMPG/FPG >270 milligram/deciliter (mg/dL) (15.0 mmol/L), from Week 8 to Week 12: fasting SMPG/FPG >240 mg/dL (13.3 mmol/L), and from Week 12 to Week 24: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c >8.5%. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline up to Week 24
Population: mITT population. The "Placebo (Two-step Titration)" and "Placebo (One-step Titration)" Arms/Groups were combined as pre-specified in the study protocol
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 159 | 160 | 160
percentage of participants | 4.4 | 3.1 | 1.3

7. Other Pre Specified Outcome: Percentage of Patients With at Least 5% Weight Loss From Baseline at Week 24
Description: as for outcome 4
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.The "Placebo (Two-step Titration)" and "Placebo (One-step Titration)" Arms/Groups were combined as pre-specified in the study protocol
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 158 | 155 | 158
percentage of participants | 15.2 | 25.8 | 19.6

8. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia and Severe Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the patient required the assistance of another person and was associated with either a plasma glucose level below 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose administration, for up to 112 weeks
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.The "Placebo (Two-step Titration)" and "Placebo (One-step Titration)" Arms/Groups were combined as pre-specified in the study protocol
Measure: Number; unit: participants
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 160 | 161 | 161
participants
  Symptomatic hypoglycemia | 12 | 12 | 6
  Severe symptomatic hypoglycemia | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 3 days after the last dose administration, for up to 112 weeks
Description: Median exposure to study treatment was 567, 588 and 589 days in lixisenatide two step titration, one step titration and placebo combined arms, respectively. The analysis was performed on safety population, defined as all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Placebo (Two-step Titration): 2-step initiation regimen of volume matching placebo.
- Placebo (One-step Titration): 1-step initiation regimen of volume matching placebo.
- Lixisenatide One-step Titration: 1-step initiation regimen of lixisenatide.
- Lixisenatide (Combined): Included all patients who received 2-step initiation regimen of lixisenatide and 1-step initiation regimen of lixisenatide.
Arm/Group | Placebo (Two-step Titration) | Placebo (One-step Titration) | Placebo (Combined) | Lixisenatide (Two-step Titration) | Lixisenatide One-step Titration | Lixisenatide (Combined)
Serious Adverse Events (participants affected / at risk) | 13/79 | 9/81 | 22/160 | 21/161 | 16/161 | 37/322
Other Adverse Events (participants affected / at risk) | 51/79 | 53/81 | 104/160 | 119/161 | 101/161 | 220/322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Two-step Titration) (N=79) | Placebo (One-step Titration) (N=81) | Placebo (Combined) (N=160) | Lixisenatide (Two-step Titration) (N=161) | Lixisenatide One-step Titration (N=161) | Lixisenatide (Combined) (N=322)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Hepatitis B (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 2
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 1
Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 2
Adams-Stokes syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 1 | 1 | 2
Bradycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Blood calcitonin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Two-step Titration) (N=79) | Placebo (One-step Titration) (N=81) | Placebo (Combined) (N=160) | Lixisenatide (Two-step Titration) (N=161) | Lixisenatide One-step Titration (N=161) | Lixisenatide (Combined) (N=322)
Bronchitis (Infections and infestations) | 6 | 7 | 13 | 3 | 7 | 10
Gastroenteritis (Infections and infestations) | 7 | 2 | 9 | 4 | 7 | 11
Influenza (Infections and infestations) | 9 | 9 | 18 | 20 | 11 | 31
Nasopharyngitis (Infections and infestations) | 13 | 8 | 21 | 16 | 18 | 34
Pharyngitis (Infections and infestations) | 6 | 6 | 12 | 9 | 10 | 19
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 9 | 4 | 6 | 10
Urinary tract infection (Infections and infestations) | 6 | 5 | 11 | 11 | 10 | 21
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 0 | 4 | 1 | 4 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 5 | 13 | 12 | 6 | 18 — Hypoglycaemia adverse event is based on investigator reported hypoglycaemia.
Dizziness (Nervous system disorders) | 11 | 10 | 21 | 19 | 15 | 34
Headache (Nervous system disorders) | 11 | 9 | 20 | 23 | 20 | 43
Hypertension (Vascular disorders) | 2 | 10 | 12 | 12 | 9 | 21
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 7 | 9 | 8 | 17
Constipation (Gastrointestinal disorders) | 3 | 0 | 3 | 11 | 2 | 13
Diarrhoea (Gastrointestinal disorders) | 10 | 11 | 21 | 24 | 16 | 40
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 7 | 9 | 16
Gastritis (Gastrointestinal disorders) | 4 | 0 | 4 | 8 | 7 | 15
Nausea (Gastrointestinal disorders) | 8 | 5 | 13 | 61 | 47 | 108
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 29 | 21 | 50
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 5 | 14 | 11 | 9 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 3 | 11 | 15 | 18 | 33
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 8 | 2 | 4 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 6 | 4 | 5 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 8 | 4 | 3 | 7
Asthenia (General disorders) | 0 | 1 | 1 | 9 | 3 | 12
Oedema peripheral (General disorders) | 4 | 3 | 7 | 3 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.